CLINICAL TRIAL: NCT06010966
Title: Effect of Intermittent TBS on Children With ADHD
Brief Title: Effect of iTBS on Children With ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hu ShaoHua, professor, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT20220110C-R2
Record Dates: First submitted 2023-07-26; First posted 2023-08-25 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-07

CONDITIONS: ADHD; rTMS
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- sham group (Sham Comparator): receive sham itbs
  Interventions: Device: rTMS
- low-dose group (Active Comparator): receive low dose of itbs
  Interventions: Device: rTMS
- high-dose group (Active Comparator): receive high dose of itbs
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — intermittent theta-burst stimulation (iTBS)

SUMMARY:
Attention Deficit/Hyperactivity Disorder (ADHD) is a common neurodevelopmental disorder characterized by persistent symptoms of attention deficit and/or hyperactivity/impulsivity . Currently, the first line drugs for treating ADHD are central stimulants such as Tomoxetine and Guanfaxine. However, there is a risk of drug abuse and misuse, which often affects sleep and appetite, only 50% of patients can fully tolerate. This project uses the iTBS stimulation on weekends, children with ADHD finish scale evaluation, magnetic resonance imaging analysis, and cognitive function before and after stimulation, This study explores its therapeutic effect on attention deficit in children and adolescents with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD in accordance with DSM-V;
* Age 6-12 years old, regardless of gender
* Right-handed
* Han nationality or born in the Han nationality Ghetto
* The course of the disease is greater than 6 months
* Webster children's intelligence ≥ 70
* The patient's guardian agrees and signs an informed consent form.

Exclusion Criteria:

* Concomitant mental disorders such as anxiety and depression;
* Widespread developmental disorders and other neurological developmental related disorders;
* Complication with other important organ diseases such as heart and lungs;
* Suffering from diseases such as epilepsy and tic disorder;
* Individuals who cannot tolerate rTMS treatment or cannot cooperate with treatment.
* Patients taking psychoactive drugs, antipsychotics, antidepressants, or mood stabilizers 3 months prior to enrollment or during rTMS treatment; In addition to the minimum effective therapeutic dose of Tomoxetine (1.2-1.4 mg • kg/day), there has been systematic use of first-line ADHD drugs in clinical practice Webster's intelligence<70
* Implantation of metal and electronic components in the body (excluding the oral cavity), such as pacemakers;

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
ADHD-RS | 4 weeks
  Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS), range from 0 to 54 points. The high scores means the worse outcome.

SECONDARY OUTCOMES:
fMRI | 4 weeks
  functional magnetic resonance imaging
Stroop color-wordtask (SCWT) | 4 weeks
  In the SCWT, the stimuli were two Chinese color words (green and red) presented in matching or contrasting font colors. The participants were asked to respond to the color of the font as quickly and as accurately as possible when a word was presented
TMT task | 4 weeks
  trailmaking test,TMT；It is divided into two parts: A and B. Part A requires the participants to connect 25 numbers on the paper in order (Figure 2). Part B includes 1-13 numbers and A-L12 letters, requiring participants to alternately connect these numbers and letters in orde

CONTACTS AND LOCATIONS:
Overall Officials: Shaohua Hu, Dr, Study Chair — Zhejiang University
Locations (1):
- Department of Psychiatry, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) is aviliable from Principal investigator